CLINICAL TRIAL: NCT03411356
Title: Comparison of Weight Loss Induced by Intermittent Fasting Versus Daily Caloric Restriction in Individuals With Obesity: A 1-Year Randomized Trial
Brief Title: Intermittent Fasting Versus Daily Caloric Restriction for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0369; R01DK111622-01A1 (NIH)
Record Dates: First submitted 2018-01-04; First posted 2018-01-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Caloric Restriction (DCR) (Active Comparator): Participants in this group will focus on daily calorie restriction as their dietary weight loss strategy.
  Interventions: Behavioral: Daily Caloric Restriction (DCR)
- Intermittent Fasting (IMF) (Experimental): Participants in this group will focus on modified intermittent fasting as their dietary weight loss strategy.
  Interventions: Behavioral: Intermittent Fasting (IMF)

INTERVENTIONS:
Behavioral: Daily Caloric Restriction (DCR) — Participants in this group will be given a calorie goal designed to produce a 34.3% energy deficit from estimated baseline weight maintenance energy requirements. Participants in this group will also receive a 12 month comprehensive group-based behavioral weight loss program and will be instructed in specific strategies to support DCR. Randomized groups will meet separately. Participants in this group will also be asked to increase moderate intensity physical activity to a target of 300 minutes per week.
  Arms: Daily Caloric Restriction (DCR)
Behavioral: Intermittent Fasting (IMF) — Participants in this group will be instructed to limit energy intake to 20% of estimated baseline energy requirements on three non-consecutive days per week, and to eat ad libitum the other 4 days per week. Participants in this group will also receive a 12 month comprehensive group based behavioral weight loss program and will be instructed in specific strategies to support IMF. Randomized groups will meet separately. Participants in this group will also be asked to increase moderate intensity physical activity to a target of 300 minutes per week.
  Arms: Intermittent Fasting (IMF)

SUMMARY:
The primary aim of this study is to is to determine if intermittent fasting (IMF) is an effective dietary strategy for treatment of obesity. A 1 year randomized trial will be used to compare weight loss generated by IMF versus Daily Caloric Restriction (DCR). The targeted weekly energy deficit is designed to be similar (~30%) and a comprehensive behavioral support program will be provided to both groups. The primary outcome is weight change at the end of the 1 year intervention; follow up measures will also be obtained 6 months after completing the intervention. This study will provide robust data regarding weight loss effectiveness of IMF and will further our understanding of the impact of IMF on energy balance.

DETAILED DESCRIPTION:
Restricting daily calorie intake is the primary dietary strategy currently used to treat obesity. However, this approach is not effective for all individuals. Further, adherence to daily caloric restriction (DCR) typically decreases over time and many individuals who lose weight with this strategy will regain. Thus, novel dietary interventions are needed to provide a broader range of treatment options. The objective of this proposal is to determine if intermittent fasting (IMF) is an effective dietary strategy for treatment of obesity. IMF is an alternative method of reducing energy intake (EI) which has gained lay popularity in recent years as a strategy for weight loss. Short-term studies suggest IMF produces 3-8% weight loss in individuals with overweight and obesity. However, few studies have compared IMF to DCR and no studies have evaluated whether IMF is an effective long-term (≥1 year) weight loss strategy. Data from an 8-week pilot study comparing IMF to DCR suggests IMF is safe, tolerable, and produces similar short-term weight loss. After 6 months of unsupervised follow-up, changes in body composition tended to be more favorable with IMF and almost twice as many IMF participants maintained a ≥5 kg weight loss. Thus, IMF may be a more effective dietary strategy for sustaining weight loss than DCR. However, longer-term data are needed and little is known about adherence to IMF or the impact of IMF on energy expenditure (EE). Short-term studies suggest adherence to IMF may be superior to DCR, however, energy intake (EI) was based on self-report which may have significant limitations. Pilot data suggests resting energy expenditure (REE) was preserved during IMF-induced weight loss, which could decrease risk for weight regain. However, the impact of IMF on other components of EE including physical activity (PA) is largely unexamined. The study design is a pragmatic randomized trial to compare weight loss generated by IMF vs DCR. The targeted weekly energy deficit will be equivalent: DCR will be prescribed a ~30% daily energy restriction and IMF will be prescribed a modified fast (~80% energy restriction) on 3 non-consecutive days per week. The hypothesis is that a weight loss program based on IMF as the primary dietary strategy will result in greater weight loss at 1 year compared to a program based on traditional DCR. The approach is innovative as the targeted energy deficit will be matched between groups and EI will be assessed objectively (using doubly-labeled water) to provide an accurate comparison of adherence. In addition, both intervention groups will receive guidelines-based behavioral support to compare IMF to the current standard of care (DCR) in a more robust fashion. This study is significant as it could identify an effective alternative dietary strategy to help more people achieve and sustain weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* Age 18-60 years
* Body Mass Index 27-46 kg/m2
* Sedentary: defined as <150 minutes per week of voluntary exercise at moderate intensity or greater and < 60 min per day of total habitual physical activity (i.e. work related, transportation related) at moderate intensity or greater, over the past 3 months.
* No self-report of acute or chronic disease (cardiovascular disease (CVD), diabetes, gastrointestinal disorders and orthopedic problems in particular)
* No plans to relocate within the next 12 months
* No plans for extended travel (> 2 weeks) within the next 12 months
* No nicotine use
* Live or work within 30 minutes of the Anschutz Health and Wellness Center (AHWC) (exceptions may be made at the discretion of the Study PI on a case by case basis for highly motivated subjects).
* Capable and willing to give informed consent, understand exclusion criteria, and accept the randomized group assignment.
* Have a primary care physician (or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
* For Females

  * Not currently pregnant or lactating
  * Not pregnant within the past 6 months
  * Not planning to become pregnant in the next 12 months;
  * Sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception

Exclusion Criteria

* Diastolic blood pressure > 100 mm of Mercury (HG) or systolic blood pressure > 160 mm HG.
* Resting heart rate >100
* Diabetes (fasting glucose ≥126 mg/dL or Glycated Hemoglobin (A1C) ≥6.5%)
* Undiagnosed hypo- or hyper-thyroidism (TSH outside of the normal range) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable.
* Hematocrit, white blood cell count or platelets significantly outside the normal reference range.
* Triglycerides > 400 mg/dL
* LDL cholesterol > 200 mg/dL
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal Premature Ventricular Contractions (PVC's), frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc (Q-T Corrected) interval > 480 msec or other significant conduction defects.
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component including: CVD, peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection, significant gastrointestinal disorders (described below), significant pulmonary disorders (described below), significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism
* Regular use of systemic steroids (other than Oral Contraceptive Pills).
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Current alcohol or substance abuse
* Nicotine use (past 6 months)
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder.
* Current severe depression or history of severe depression within the previous year, based on Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria for Major Depressive Episode.
* History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary or exercise interventions.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials.
* Weight loss >5kg in past 3 months for any reason except post-partum weight loss, weight gain >5kg in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline and weeks 4, 13, 26, 39, 52.
  Body weight will be measured via clinic scale.

SECONDARY OUTCOMES:
Change in Body Weight | Week 78.
  Body weight will be measured via clinic scale. The 78 month time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up weight.
Changes in Body Composition | Baseline and weeks 26, 52, and 78.
  Body composition will be assessed with dual-energy x-ray absorptiometry (DXA).The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Blood Pressure | Baseline and weeks 13, 26, 52, and 78.
  Blood pressure will be measured with a sphygomanometer. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Fasting Lipids | Baseline and weeks 26, 52, and 78.
  12 hour fasting blood sample for measurement of lipid profile.The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Insulin Sensitivity | Baseline and weeks 26, 52, and 78.
  12 hour fasting blood sample for measurement of insulin and glucose. Insulin sensitivity (homeostasis model assessment of insulin resistance [HOMA-IR]) will be calculated as ([insulin] x [fasting glucose x 0.055]/22.5). The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Objectively Measured Energy Intake (EI) | Baseline, weeks 26, 52, and 78.
  EI will be measured using the doubly-labeled water (DLW) intake-balance method. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Self-Reported Energy Intake (EI) | Baseline and weeks 13, 26, 52, and 78.
  Dietary energy intake (kcals/day) will be measured with diet diaries. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Self-reported Diet Composition | Baseline and weeks 13, 26, 52, and 78.
  Dietary macronutrient intake will be measured with diet diaries. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Self-Reported Dietary Adherence | Weeks 4, 8, 13, 18, 22, 26, 30, 34, 39, 44, 48, 52
  Adherence to prescribed diet will be assessed with a monthly questionnaire.
Changes in Resting Energy Expenditure (REE) | Baseline and weeks 26, 52, and 78.
  REE will be measured using indirect calorimetry. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Total Daily Energy Expenditure (TDEE) | Baseline and weeks 26, 52, and 78.
  TDEE will be measured using the doubly-labeled water (DLW) method. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Physical Activity | Baseline and weeks 13, 26, 52, and 78.
  Physical activity will be measured with activity monitors. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.
Changes in Sedentary Behavior | Baseline and weeks 13, 26, 52, and 78.
  Sedentary behavior will be measured with activity monitors. The 78 week time point was added via a protocol amendment after study start. This is not a primary outcome, but rather a 6-month post-primary outcome follow-up measure.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Catenacci, MD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- Kristen Bing, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Breit MJ, Pan Z, Ostendorf DM, Dahle JH, Catenacci VA, Creasy SA, Melanson EL. Using Time-Weighted Averages of Total Daily Energy Expenditure to Estimate Energy Intake During a Weight Loss Intervention. Obesity (Silver Spring). 2025 Nov;33(11):2093-2102. doi: 10.1002/oby.70008. Epub 2025 Aug 28. PMID 40878019
- [Derived] Catenacci VA, Ostendorf DM, Pan Z, Kaizer LK, Creasy SA, Zaman A, Caldwell AE, Dahle J, Swanson B, Breit MJ, Bing K, Wayland LT, Panter SL, Scorsone JJ, Bessesen DH, MacLean P, Melanson EL. The Effect of 4:3 Intermittent Fasting on Weight Loss at 12 Months : A Randomized Clinical Trial. Ann Intern Med. 2025 May;178(5):634-644. doi: 10.7326/ANNALS-24-01631. Epub 2025 Apr 1. PMID 40163873